CLINICAL TRIAL: NCT02561819
Title: Measurement of Body Composition by Air Displacement Plethysmography in Pediatric Intestinal Failure Patients
Status: Completed | Type: Observational
Sponsor: Christopher Duggan (Other)
Responsible Party: Sponsor-Investigator, Christopher Duggan, MD, MPH, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Other Study IDs: IRB-P00014026
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; Congenital Short Bowel Syndrome; Body Composition; Parenteral Nutrition; Intestinal Failure
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Pseudo-Obstruction; Hyperphagia; Intestinal Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will determine if air-displacement plethysmography (ADP) provides accurate measurement of body composition (percent body fat and fat-free mass) in pediatric patients with intestinal failure, as compared to body composition measured by alternative standard methods, including deuterium dilution, bioimpedance analysis (BIA), dual x-ray absorptiometry (DXA) when clinically indicated, and routine anthropometric measurements.

DETAILED DESCRIPTION:
Infants and children with intestinal failure (IF) require prolonged periods of parenteral nutrition (PN) for sustenance and growth until intestinal adaptation allows adequate enteral intake. Lean body mass (or muscle mass) preservation and accrual is an important goal during this phase of nutritional rehabilitation. However, lean body mass is not accurately measured by currently available anthropometric techniques. Thus, despite weight gain, muscle mass depletion can remain undetected.

Little data exist in the field of measuring body composition in patients with intestinal failure, where changes in body weight are commonly taken to indirectly measure gastrointestinal absorptive function. Body composition analysis is of particular importance in the management of these patients, since it can help guide medical, surgical and/or nutrition interventions, including titration of enteral or parenteral nutrition. To the investigators' knowledge there are no studies examining whether air-displacement plethysmography (ADP) is a valid measure of body composition in patients with intestinal failure.

The investigators propose a non-randomized, prospective cohort study to validate ADP as a measure of body composition in infants and children with IF.

The investigators will apply non-radioactive (stable) isotope techniques to examine the accuracy of ADP in measuring body composition in these children.

The investigators will also compare ADP with bioimpedance analysis and routine anthropometry. Additionally, if subjects have had a recent dual-energy X- ray absorptiometry (DXA) scan, the investigators will compare the ADP estimates of body composition to those obtained from DXA. The investigators hypothesize that ADP is a feasible and accurate technique for body composition measurements, and that the device can be used to serially measure lean body mass and fat mass changes in this cohort. If the feasibility and accuracy of ADP for body composition analysis can be demonstrated, the technique is likely to have wider applications in other pediatric illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated in the CAIR Program at Boston Children's Hospital will be eligible for participation if they meet the definition of short bowel syndrome and are under 18 years of age. Short bowel syndrome will be defined as a malabsorptive state resulting from congenital or acquired gastrointestinal disease leading to current dependence on parenteral nutrition for greater than or equal to 90 days. If the patient is on intravenous fluids, they must have a stable intravenous fluid regimen for at least 4 weeks prior to the study visit.

Exclusion Criteria:

* age < 2 years or ≥ 18 years
* presence of cardiac pacing device (BIA may theoretically interfere with pacer functioning)
* presence of any other electrical device that might interfere with the BIA such as implantable drug delivery pumps, vagal nerve stimulator and invasive cerebral perfusion monitor
* subjects will be excluded due to pregnancy
* subjects with ongoing fluid imbalance, clinically evident shifts in fluid compartments (e.g. edema, ascites) or with fluid resuscitation (defined as daily fluid intake more than 150% of maintenance or fluid boluses more than 20 ml/kg/day). Determination of fluid imbalance will be made by the physicians directly involved in the patient's care.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with intestinal failure between 2-17 years of age inclusive will be recruited through the Center for Advanced Intestinal Rehabilitation (CAIR) program at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-12

PRIMARY OUTCOMES:
Body composition (percent body fat and fat-free mass) as measured by air displacement plethysmography in pediatric patients with intestinal failure on date of visit. | Single Visit
  Body composition (percent body fat and fat-free mass) as measured by air displacement plethysmography in pediatric patients with intestinal failure will be compared to body composition measurements done by the deuterium dilution technique, DXA scan, and bioimpedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Duggan, MD, MPH, Principal Investigator — Boston Children's Hospital; Alexandra Carey, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Keefe SJ, Buchman AL, Fishbein TM, Jeejeebhoy KN, Jeppesen PB, Shaffer J. Short bowel syndrome and intestinal failure: consensus definitions and overview. Clin Gastroenterol Hepatol. 2006 Jan;4(1):6-10. doi: 10.1016/j.cgh.2005.10.002. PMID 16431298
- [Background] Gosselin KB, Duggan C. Enteral nutrition in the management of pediatric intestinal failure. J Pediatr. 2014 Dec;165(6):1085-90. doi: 10.1016/j.jpeds.2014.08.012. Epub 2014 Sep 18. No abstract available. PMID 25242686
- [Background] Winkler MF, Smith CE. Clinical, social, and economic impacts of home parenteral nutrition dependence in short bowel syndrome. JPEN J Parenter Enteral Nutr. 2014 May;38(1 Suppl):32S-37S. doi: 10.1177/0148607113517717. Epub 2014 Jan 13. PMID 24418898
- [Background] Squires RH, Duggan C, Teitelbaum DH, Wales PW, Balint J, Venick R, Rhee S, Sudan D, Mercer D, Martinez JA, Carter BA, Soden J, Horslen S, Rudolph JA, Kocoshis S, Superina R, Lawlor S, Haller T, Kurs-Lasky M, Belle SH; Pediatric Intestinal Failure Consortium. Natural history of pediatric intestinal failure: initial report from the Pediatric Intestinal Failure Consortium. J Pediatr. 2012 Oct;161(4):723-8.e2. doi: 10.1016/j.jpeds.2012.03.062. Epub 2012 May 11. PMID 22578586
- [Background] Sharma TS, Bechard LJ, Feldman HA, Venick R, Gura K, Gordon CM, Sonis A, Guinan EC, Duggan C. Effect of titrated parenteral nutrition on body composition after allogeneic hematopoietic stem cell transplantation in children: a double-blind, randomized, multicenter trial. Am J Clin Nutr. 2012 Feb;95(2):342-51. doi: 10.3945/ajcn.111.026005. Epub 2011 Dec 28. PMID 22205317
- [Background] Murphy AJ, Wells JC, Williams JE, Fewtrell MS, Davies PS, Webb DK. Body composition in children in remission from acute lymphoblastic leukemia. Am J Clin Nutr. 2006 Jan;83(1):70-4. doi: 10.1093/ajcn/83.1.70. PMID 16400052
- [Background] Burnham JM, Shults J, Semeao E, Foster BJ, Zemel BS, Stallings VA, Leonard MB. Body-composition alterations consistent with cachexia in children and young adults with Crohn disease. Am J Clin Nutr. 2005 Aug;82(2):413-20. doi: 10.1093/ajcn.82.2.413. PMID 16087987
- [Background] Stallings VA, Tomezsko JL, Schall JI, Mascarenhas MR, Stettler N, Scanlin TF, Zemel BS. Adolescent development and energy expenditure in females with cystic fibrosis. Clin Nutr. 2005 Oct;24(5):737-45. doi: 10.1016/j.clnu.2005.02.005. Epub 2005 Apr 8. PMID 16182037
- [Background] Farrell AG, Schamberger MS, Olson IL, Leitch CA. Large left-to-right shunts and congestive heart failure increase total energy expenditure in infants with ventricular septal defect. Am J Cardiol. 2001 May 1;87(9):1128-31, A10. doi: 10.1016/s0002-9149(01)01479-5. No abstract available. PMID 11348620
- [Background] Ellis KJ, Shypailo RJ, Wong WW. Measurement of body water by multifrequency bioelectrical impedance spectroscopy in a multiethnic pediatric population. Am J Clin Nutr. 1999 Nov;70(5):847-53. doi: 10.1093/ajcn/70.5.847. PMID 10539745
- [Background] Elberg J, McDuffie JR, Sebring NG, Salaita C, Keil M, Robotham D, Reynolds JC, Yanovski JA. Comparison of methods to assess change in children's body composition. Am J Clin Nutr. 2004 Jul;80(1):64-9. doi: 10.1093/ajcn/80.1.64. PMID 15213029
- [Background] Ginde SR, Geliebter A, Rubiano F, Silva AM, Wang J, Heshka S, Heymsfield SB. Air displacement plethysmography: validation in overweight and obese subjects. Obes Res. 2005 Jul;13(7):1232-7. doi: 10.1038/oby.2005.146. PMID 16076993
- [Background] Gately PJ, Radley D, Cooke CB, Carroll S, Oldroyd B, Truscott JG, Coward WA, Wright A. Comparison of body composition methods in overweight and obese children. J Appl Physiol (1985). 2003 Nov;95(5):2039-46. doi: 10.1152/japplphysiol.00377.2003. PMID 14555670
- [Background] Schoeller DA, van Santen E, Peterson DW, Dietz W, Jaspan J, Klein PD. Total body water measurement in humans with 18O and 2H labeled water. Am J Clin Nutr. 1980 Dec;33(12):2686-93. doi: 10.1093/ajcn/33.12.2686. PMID 6776801
- [Background] Van Kreel BK, Van der Vegt F, Meers M, Wagenmakers T, Westerterp K, Coward A. Determination of total body water by a simple and rapid mass spectrometric method. J Mass Spectrom. 1996 Jan;31(1):108-11. doi: 10.1002/(SICI)1096-9888(199601)31:13.0.CO;2-M. PMID 8799264
- [Background] Wong WW, Cochran WJ, Klish WJ, Smith EO, Lee LS, Klein PD. In vivo isotope-fractionation factors and the measurement of deuterium- and oxygen-18-dilution spaces from plasma, urine, saliva, respiratory water vapor, and carbon dioxide. Am J Clin Nutr. 1988 Jan;47(1):1-6. doi: 10.1093/ajcn/47.1.1. PMID 3122550
- [Background] Andersen GS, Girma T, Wells JC, Kaestel P, Leventi M, Hother AL, Michaelsen KF, Friis H. Body composition from birth to 6 mo of age in Ethiopian infants: reference data obtained by air-displacement plethysmography. Am J Clin Nutr. 2013 Oct;98(4):885-94. doi: 10.3945/ajcn.113.063032. Epub 2013 Aug 28. PMID 23985805
- [Background] Plasqui G, Soenen S, Westerterp-Plantenga MS, Westerterp KR. Measurement of longitudinal changes in body composition during weight loss and maintenance in overweight and obese subjects using air-displacement plethysmography in comparison with the deuterium dilution technique. Int J Obes (Lond). 2011 Aug;35(8):1124-30. doi: 10.1038/ijo.2010.250. Epub 2010 Nov 23. PMID 21102553
- [Background] Rosendale RP, Bartok CJ. Air-displacement plethysmography for the measurement of body composition in children aged 6-48 months. Pediatr Res. 2012 Mar;71(3):299-304. doi: 10.1038/pr.2011.42. Epub 2012 Jan 18. PMID 22258086
- [Background] Prior BM, Cureton KJ, Modlesky CM, Evans EM, Sloniger MA, Saunders M, Lewis RD. In vivo validation of whole body composition estimates from dual-energy X-ray absorptiometry. J Appl Physiol (1985). 1997 Aug;83(2):623-30. doi: 10.1152/jappl.1997.83.2.623. PMID 9262461
- [Background] Buchholz AC, Bartok C, Schoeller DA. The validity of bioelectrical impedance models in clinical populations. Nutr Clin Pract. 2004 Oct;19(5):433-46. doi: 10.1177/0115426504019005433. PMID 16215137
- [Background] Bunt JC, Lohman TG, Boileau RA. Impact of total body water fluctuations on estimation of body fat from body density. Med Sci Sports Exerc. 1989 Feb;21(1):96-100. doi: 10.1249/00005768-198902000-00017. PMID 2927308
- [Background] Mehta NM, Raphael B, Guteirrez IM, Quinn N, Mitchell PD, Litman HJ, Jaksic T, Duggan CP. Comparison of body composition assessment methods in pediatric intestinal failure. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):99-105. doi: 10.1097/MPG.0000000000000364. PMID 24614122
- [Background] Zemel BS, Riley EM, Stallings VA. Evaluation of methodology for nutritional assessment in children: anthropometry, body composition, and energy expenditure. Annu Rev Nutr. 1997;17:211-35. doi: 10.1146/annurev.nutr.17.1.211. PMID 9240926
- [Background] Pichler J, Chomtho S, Fewtrell M, Macdonald S, Hill SM. Growth and bone health in pediatric intestinal failure patients receiving long-term parenteral nutrition. Am J Clin Nutr. 2013 Jun;97(6):1260-9. doi: 10.3945/ajcn.112.057935. Epub 2013 Apr 10. PMID 23576042
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Goulet O, Baglin-Gobet S, Talbotec C, Fourcade L, Colomb V, Sauvat F, Jais JP, Michel JL, Jan D, Ricour C. Outcome and long-term growth after extensive small bowel resection in the neonatal period: a survey of 87 children. Eur J Pediatr Surg. 2005 Apr;15(2):95-101. doi: 10.1055/s-2004-821214. PMID 15877257